CLINICAL TRIAL: NCT02059200
Title: The Effectiveness of Mindfulness Based Compassionate Living in Recurrent Depression
Brief Title: Mindfulness Based Compassionate Living in Recurrent Depression
Acronym: MBCL-RD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Triodos Foundation (Unknown)
Responsible Party: Principal Investigator, Anne Speckens, Professor, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MFN-MBCL-2013-2017
Record Dates: First submitted 2014-01-30; First posted 2014-02-11 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Recurrent Depression
Keywords: Randomised controlled trial; Recurrent depression; Mindfulness training; Compassion training (MBCL); Fear of Compassion; Added value Compassion
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MBCL + TAU (Experimental): This cohort receives the Mindfulness Based Compassionate Living program in addition to treatment as usual.
  Interventions: Behavioral: Mindfulness Based Compassionate Living
- TAU (No Intervention): This cohort receives treatment as usual of any nature, e.g. psychotherapy, antidepressant medication etc.

INTERVENTIONS:
Behavioral: Mindfulness Based Compassionate Living — The MBCL program consists of eight biweekly group sessions of 2.5 hours, in which the participants get formal meditation exercises, some theoretical information and participate in inquiry on the meditation exercises and homework assignments. Homework assignments are given after every session, consisting of formal and informal meditation exercises primarily and some diary instructions.
  Other Names: MBCL; Mindfulness Based Compassion Training
  Arms: MBCL + TAU

SUMMARY:
Since a few years, Mindfulness Based Cognitive Therapy (MBCT) has been used as treatment for patients suffering from recurrent depression. Though a number of studies show that MBCT is effective in this population and MBCT reduces the chances of relapse/recurrence in recurrent depressive patients, the chance of a new depression developing after end of treatment is still considerable. Ergo, there is room for improvement.

Especially the development of a non-judging or compassionate attitude towards all experience seems to mediate the treatment effect. It is therefore our expectation that a follow-up intervention that focuses specifically on self-compassion could prove very useful in elaborating on the effects of MBCT.

The research question of this research is therefore: what is the effect of compassion training in people suffering from recurrent depression who have already received MBCT training?

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent depression according to the DSM-IV criteria.
2. Having participated in an MBCT training (>= 4 sessions)

Exclusion Criteria:

1. One or more previous (hypo)manic episodes according to DSM-IV criteria.
2. Primary psychotic disorder, e.g. schizophrenia or delusions.
3. Clinically relevant neurological conditions (e.g. brain trauma or dementia) or somatic conditions (e.g. cancer, AIDS) that could be related to the depression.
4. Current alcohol and/or drug abuse.
5. Use of high dosages of benzodiazepines.
6. Recent electro convulsive therapy (ECT) (less than 3 months ago).
7. Problems impeding participating in a group, such as severe borderline personality disorder.
8. No prior experience with MBCT.
9. Problems impeding completing the questionnaires, such as cognitive dysfunctions (only assessed if suspected).
10. Subnormal intelligence (IQ < 80) (only assessed if suspected).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II | 1 year
  The BDI-II measures depression symptoms. Measurements will be taken at baseline, end of treatment/control and follow up.

SECONDARY OUTCOMES:
Self-Compassion Scale | 1 year
  The Self-Compassion Scale measures Self-Compassion. Measurements will be taken at baseline, end of treatment/control and follow-up.
Five Facet Mindfulness Questionnaire | 1 year
  The FFMQ measures mindfulness skills. Measurements will be taken at baseline, end of treatment/control and follow-up.
The Acceptance and Action Questionnaire-II | 1 year
  The AAQ-II measures Experiential Avoidance. Measurements will be taken at baseline, end of treatment/control and follow-up.
Fears of Compassion Scale (3) | 1 year
  The FoCS (3) measures fear of Self-Compassion. Measurements will be taken at baseline, end of treatment/control and follow-up.
Types of Positive Affect Scale | 1 year
  The TPAS measures Positive Affect. Measurements will be taken at baseline, end of treatment/control and follow-up.
The World Health Organization Quality of Life Scale | 1 year
  The WHO-QoL measures Quality of Life. Measurements will be taken at baseline, end of treatment/control and follow-up.
The Ruminative Response Scale | 1 year
  The RRS measures Rumination. Measurements will be taken at baseline, end of treatment/control and follow-up.
The Childhood Trauma Questionnaire | Baseline
  The CTQ measures Childhood Adversity. Measurements will be taken at baseline only.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Speckens, Professor, Principal Investigator — University Medical Center Nijmegen
Locations (1):
- University Medical Center Nijmegen, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Schuling R, Huijbers MJ, van Ravesteijn H, Donders R, Cillessen L, Kuyken W, Speckens AEM. Recovery from recurrent depression: Randomized controlled trial of the efficacy of mindfulness-based compassionate living compared with treatment-as-usual on depressive symptoms and its consolidation at longer term follow-up. J Affect Disord. 2020 Aug 1;273:265-273. doi: 10.1016/j.jad.2020.03.182. Epub 2020 May 4. PMID 32421612
- [Derived] Schuling R, Huijbers MJ, van Ravesteijn H, Donders R, Kuyken W, Speckens AE. A parallel-group, randomized controlled trial into the effectiveness of Mindfulness-Based Compassionate Living (MBCL) compared to treatment-as-usual in recurrent depression: Trial design and protocol. Contemp Clin Trials. 2016 Sep;50:77-83. doi: 10.1016/j.cct.2016.07.014. Epub 2016 Jul 21. PMID 27451354
- See also: Related info — http://www.radboudcentrumvoormindfulness.nl